CLINICAL TRIAL: NCT05360043
Title: Efficacy and Safety of 1565-nm Non-ablative Fractional Laser Versus Long-pulsed 1064-nm Nd:YAG Laser in the Treatment of Enlarged Facial Pores
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-0073
Record Dates: First submitted 2022-04-06; First posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Enlarged Facial Pores
Keywords: Facial pores; Non-ablative fractional laser; Long-pulsed Nd:YAG laser
MeSH Terms: interventions — Laser Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LPNY side (Experimental): 1064-nm LPNY (Gentle YAG, Candela ®, USA)
  Interventions: Device: laser treatment
- NAFL side (Experimental): 1565-nm NAFL(ResurFX mode, M22, Lumenis ®, Yokneam, Israel)
  Interventions: Device: laser treatment

INTERVENTIONS:
Device: laser treatment — All subjects were treated with a 1565-nm NAFL on their left faces for one pass, A 34-40 mJ per microbeam laser was used, and density was 250-300 microbeam per cm2. Their right faces were treated with a 1064-nm LPNY for one pass. We used a spot size of 10 mm in diameter, an energy density of 45-50 J/cm2, pulse width of 300 microseconds, and a repetition rate of 2 Hz. 1064-nm LPNY was equipped with a dynamic cooling device (DCD), the parameter was set as 40/20/0 ms. A total of 5 treatments were carried out at 2-week intervals, and one follow-up session at two months after last treatment. Before each treatment, subjects were asked to wash their face with clean water, and no topical lotion was applied. For post-treatment care, all subjects were advised to use their own moisturizing cream and avoid sun exposure.

SUMMARY:
Facial pores are visible openings of pilosebaceous follicles, it is one of the important factors that affect the appearance of facial skin. This study aims to evaluate and compare the Efficacy and safety of 1565 nm non-ablative fractional laser (NAFL) and long-pulsed 1064 nm Nd:YAG laser (LPNY) in the treatment of enlarged facial pores.

DETAILED DESCRIPTION:
Facial pores are visible openings of pilosebaceous follicles. These openings are not fixed structures and they can be affected by many factors, including sebum secretion, skin elasticity, hair thickness, age, hormones and ultraviolet exposure. These enlarged pores remain a cosmetic problem that impacts patient quality of life. At present, there is no unified evaluation standard for enlarged facial pores, and the mechanisms that underline enlarged facial pores remain unclear.

Various methods have been used to treat enlarged facial pores mainly focus on the possible causes. Treatment options include topical retinoic acid, oral isotretinoin, antiandrogen therapy, injections of botulinum toxin type A, chemical peeling, lasers, radiofrequency, and ultrasound devices. In recent years, various studies on laser treatments of facial pores are gradually increasing because of good efficacy and limited adverse reactions.

The 1064-nm LPNY has been widely used for facial rejuvenation. Many studies have confirmed that LPNY can reduce facial wrinkles and improve skin elasticity. Some researchers have used it to treat enlarged pores, and it has shown good results. Recently, 1565-nm NAFL is introduced for skin resurfacing, it has also been shown to be effective in treating enlarged facial pores. However, there are not enough clinical researches to confirm their efficacy, and no study has compared these two laser treatments before. So this is the first self-comparative study to compare the safety and efficacy of two lasers in the treatment of enlarged facial pores.

ELIGIBILITY:
Inclusion Criteria:

* subjects with enlarged facial pores who were screened by a designated dermatologist

Exclusion Criteria:

* infectious skin disease or systemic disease; skin tumors; pregnancy and lactation; patients with a history of glucocorticoids, immunosuppressant drugs and other drugs within 4 weeks; a history of keloid; a medical history of chemical peelings, filler injections, plastic surgery, or laser therapy on the face in the last 3 months

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Estimated)
Dates: Start 2018-10-27 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Pore number | from baseline(T0) at two months after last treatment(T1)
  The VISIA Complexion Analysis System was used to take photos of both facial sides. The system can automatically measure the number of pores. When pore size is smaller or less visible, the system will not detect it, and the pore count will be lower.
Subjective evaluations for improvement in appearance of facial pores | two months after last treatment(T1)
  Subjects were asked to evaluate the improvement of pore appearance after each treatment and follow-up, rated on a 4-point grading scale. 0=No significant change (0-10%); 1=Mild improvement (11-25%); 2=Moderate improvement (26-50%); 3=Marked improvement (51-75%); 4=Very significant improvement (76-100%).
Satisfaction evaluations for treatment results | two months after last treatment(T1)
  Subjects rated their satisfaction with the treatment results, using a Likert satisfaction scale (1-5). 1=Very dissatisfied; 2=Dissatisfied; 3=Neither satisfied nor dissatisfied; 4=Satisfied; 5=Very satisfied.

SECONDARY OUTCOMES:
Pain score | immediately after each laser treatment
  Subjects were asked to rate the degree of pain post-treatment using a numerical rating scale (NRS) ranging from 0 (no pain) to 10 (unbearable pain).
Side effects | through study completion, an average of 0.5 year
  Any side effects or complications were recorded at each visit, including erythema, edema, and pigmentation, et al.

CONTACTS AND LOCATIONS:
Overall Officials: Suiqing Cai, Ph.D, Study Director — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital of Zhejiang University of Medicine, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang Y, Zheng Y, Cai S. Efficacy and safety of 1565-nm non-ablative fractional laser versus long-pulsed 1064-nm Nd:YAG laser in treating enlarged facial pores. Lasers Med Sci. 2022 Oct;37(8):3279-3284. doi: 10.1007/s10103-022-03622-z. Epub 2022 Aug 15. PMID 35971017